CLINICAL TRIAL: NCT02235831
Title: DAILIES® AquaComfort Plus® MF - Comparative Assessment of Visual Performance Using Objective Measurements
Brief Title: DAILIES® AquaComfort Plus® Multifocal (MF) - Comparative Assessment of Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLT330-P001
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Presbyopia; Refractive Error
Keywords: DACP MF; DAILIES AquaComfort Plus® Multifocal; presbyopia; visual performance
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DACP MF (Experimental): DACP MF worn first, followed by DACP and DACP MF (Low Add) as randomized. Lenses worn for 5±1 days, 6 hours per day, in a daily wear daily disposable modality. DACP MF will be worn bilaterally (in both eyes).
  Interventions: Device: Nelfilcon A MF contact lenses (DACP MF); Device: Nelfilcon A single vision contact lenses (DACP)
- DACP (Active Comparator): DACP worn first, followed by DACP MF and DACP MF (Low Add), as randomized. Lenses worn for 5±1 days, 6 hours per day, in a daily wear daily disposable modality. DACP worn as monovision (distance correction in one eye and near correction in the other eye).
  Interventions: Device: Nelfilcon A MF contact lenses (DACP MF); Device: Nelfilcon A single vision contact lenses (DACP)
- DACP MF (Low Add) (Active Comparator): DACP MF (Low Add) worn first, followed by DACP and DACP MF, as randomized. Lenses worn for 5±1 days, 6 hours per day, in a daily wear daily disposable modality. DACP MF (Low Add) worn bilaterally (in both eyes).
  Interventions: Device: Nelfilcon A MF contact lenses (DACP MF); Device: Nelfilcon A single vision contact lenses (DACP)

INTERVENTIONS:
Device: Nelfilcon A MF contact lenses (DACP MF) — Multifocal contact lenses in Low, Medium, High Add
Device: Nelfilcon A single vision contact lenses (DACP)

SUMMARY:
The purpose of this study is to evaluate the visual performance of DAILIES® Aqua Comfort Plus® (DACP) MF contact lens using new objective measurements.

DETAILED DESCRIPTION:
In this 3-treatment, 3-period, 6-sequence crossover study, each subject received all 3 products in randomized order and used 1 product at a time for a duration of 5±1 days before switching to the next assigned product.

ELIGIBILITY:
Inclusion Criteria:

* History of soft contact lens wear (hydrogel or silicone hydrogel) in both eyes during the past 3 months and able to wear lenses at least 8 hours a day, 5 days a week
* Spectacle add between +1.50 and +2.50 diopters (D) (inclusive)
* Requiring lenses within the power range of both study contact lenses to be fitted
* Cylinder, if present, less or equal to 0.50D in both eyes at Visit 1
* Vision correctable to 20/30 (0.2 logMAR) or better in each eye at distance
* Acceptable fit with both study contact lenses
* Willing to wear lenses every day or at least for a minimum of 5 days per week 6 hours per day, every day if possible
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Current multifocal contact lens wearer
* Current monovision wearer or failed attempt with monovision
* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear
* Use of systemic or ocular medications which contact lens wear could be contraindicated as determined by the investigator
* Eye injury or surgery within 12 weeks immediately prior to enrollment in this trial
* Any moderate or severe ocular condition observed during the slitlamp examination at the enrollment visit
* History of herpetic keratitis, ocular surgery or irregular cornea
* Prior refractive surgery (e.g. LASIK, PRK, etc)
* Monocular (only 1 eye with functional vision) or fit with only 1 lens
* Habitually uncorrected anisometropia >2.00D
* Clinically significant anisocoria
* Participation in any clinical trial within 30 days of the enrollment visit
* Other protocol-defined exclusion criteria may apply

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, EMEA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in Spain.
Pre-assignment Details: Twenty-four subjects were enrolled; all enrolled subjects were also randomized. This reporting group includes all randomized subjects (24).
Groups:
- Seq I: DACP MF lenses worn first, followed by DACP MF (Low Add) lenses next, and DACP (monovision) lenses last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
- Seq 2: DACP MF lenses worn first, followed by DACP (monovision) lenses next, and DACP MF (Low Add) lenses last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
- Seq 3: DACP MF (Low Add) lenses worn first, followed by DACP MF lenses next, and DACP (monovision) lenses last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
- Seq 4: DACP MF (Low Add) lenses worn first, followed by DACP (monovision) lenses next, and DACP MF last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
- Seq 5: DACP (monovision) lenses first, followed by DACP MF lenses next, and DACP MF (Low Add) lenses last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
- Seq 6: DACP (monovision) lenses first, followed by DACP MF (Low Add) lenses next, and DACP MF lenses last. All lenses worn for 5±1 days in a daily wear daily disposable modality.
Period: Period 1, First 5 Days of Wear
Arm/Group | Seq I | Seq 2 | Seq 3 | Seq 4 | Seq 5 | Seq 6
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Second 5 Days of Wear
Arm/Group | Seq I | Seq 2 | Seq 3 | Seq 4 | Seq 5 | Seq 6
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3, Third 5 Days of Wear
Arm/Group | Seq I | Seq 2 | Seq 3 | Seq 4 | Seq 5 | Seq 6
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any investigational product evaluated in this study.
Groups:
- Overall: DACP MF, DACP MF (Low Add), and DACP (monovision) lenses worn in 6 different sequences as randomized in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (4.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Area for Each Region (Near and Intermediate) Under the Mean Defocus Curve (AUC) at High Luminance
Description: Visual acuity was measured with contact lenses in place using an Early Treatment Diabetic Retinopathy Study (ETDRS) high contrast logMAR chart under well-lit conditions. Lenses of different spherical powers (+2.00 diopter to -5.00 diopter) were placed in front of the eyes to produce varying levels of defocus, and logMAR acuity at each defocus value was recorded. The area under the defocus curve (AUC) was calculated via the trapezoidal rule for the entire study population by treatment using a 0.3 logMAR threshold for intermediate from -2.00 D (50cm) to -0.50 D (2m) and near from -4.00 D (25cm) to -2.00 D (50cm). A higher value indicates a bigger area of focus. This outcome measure was prespecified for monovision and DACP MF.
Time Frame: Day 5, each product
Population: This analysis population includes all randomized subjects excluding those who met the critical deviation criteria, as specified in the Deviations and Evaluability Plan (DEP).
Measure: Number; unit: diopter*logMar
Groups:
- Monovision: Nelfilcon A contact lenses worn as monovision during Period 1, 2, or 3 for 5±1 days.
- DACP MF: Nelfilcon A multifocal contact lenses worn during Period 1, 2, or 3 for 5±1 days.
Arm/Group | Monovision | DACP MF
Number analyzed (Participants) | 24 | 24
diopter*logMar
  Near | 0.09 | 0.18
  Intermediate | 0.24 | 0.36

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 19 days). This analysis group includes all subjects exposed to any investigational product evaluated in this study, based on treatment-specific exposure.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. AEs were reported by the subject or observed by the investigator.
Groups:
- DACP MF (Low Add): Nelfilcon A multifocal contact lenses worn during Period 1, 2, or 3 for 5±1 days.
Arm/Group | Monovision | DACP MF | DACP MF (Low Add)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.